CLINICAL TRIAL: NCT05194943
Title: Trends and Safety in Revisional Bariatric Surgery in Italy: a High Volume Multicenter, Observational Longitudinal Study (RBST)
Brief Title: Trends and Safety in Revisional Bariatric Surgery in Italy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, Prof, University of Roma La Sapienza
Other Study IDs: RBST2021
Record Dates: First submitted 2022-01-05; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Remission; Complication,Postoperative; Complication of Surgical Procedure; Safety Issues
Keywords: revisional bariatric surgery; safety bariatric surgery; insufficient weight loss; weight regain; gastroesophageal reflux
MeSH Terms: conditions — Obesity, Morbid; Postoperative Complications; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- 1. UOC Chirurgia Bariatrica, Policlinico San Marco, Zingonia, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 2. UOC di Chirurgia Bariatrica e Metabolica, Azienda Ospedaliera Universitaria Pisana, Pisa, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 3. UOSD Week Surgery, Chirurgia Bariatrica, Azienda Ospedale-Università di Padova, Padova, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 4. Unita di Chirurgia dell'Obesità e Metabolica, Azienda Ospedaliero-Universitaria, Bologna, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 5. UO Chirurgia Generale, Policlinico San Marco di Zingonia, Zingonia, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 6. UOC Chirurgia Bariatrica e Metabolica, Ospedale San Carlo di Nancy , Roma, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 7. Dipartimento di Scienze Chirurgiche, Azienda Ospedaliera Universitaria, Torino, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 8. UO di Chirurgia Bariatrica, Humanitas Research Hospital, Rozzano, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 9. UOC Chirurgia Generale & Bariatric Center of Excellence IFSO-EC, Latina, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 10. UOC Chirurgia Generale, Ospedale Villa d'Agri, Potenza, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures
- 11. UOC di Chirurgia Generale e d'Urgenza, Presidio Ospedaliero ARNAS, Catania, Italy: All patients undergoing revisional bariatric surgery in this center from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering reasons for surgery, technique, mortality, intraoperative and perioperative complications, readmission for any reason, following the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days.
  Interventions: Procedure: revisional bariatric surgical procedures

INTERVENTIONS:
Procedure: revisional bariatric surgical procedures — Any procedure performed as a second or third after an initial, primary bariatric surgery, performed due to complications or due to scarce results in term of weight loss and comorbidities improvement

SUMMARY:
Background: Revisional bariatric surgery (RBS) represents a further solution for patients who experience an inadequate response following initial bariatric surgery or significant weight regain following an initial satisfactory response. Studies including the follow-up of patients with complications after RBS are still lacking. Aim: to analyze the trend, mortality, and complications at 30 days after RBS in Italy. Secondary aim: 30-day readmission rate, reoperations for any reason related to bariatric surgery. Design: longitudinal, prospective, multicenter study. Time interval: 10 months October 2021 - July 2022). Setting: 11 high-volume bariatric centers of the Italian National Health Service (SSN), university hospitals, hospitals, accredited private centers. Methods: All patients undergoing RBS from 01.11.2021 through 31.04.2022 will be enrolled in a prospective, online database, registering indications, technique, mortality, intraoperative and perioperative complications, readmission for any reason. All participating centers follow the same preoperative work-up protocol, indications, informed consent, and postoperative follow-up, including scheduled telephone and outpatient visits after 7, 15 and 30 postoperative days. Inclusion criteria: revisional procedures; no concomitant procedure, but hiatal hernia repair; age >18<60 years; compensated comorbidities; informed consent including COVID-19 addendum; adherence to specific admission, in-hospital and follow-up protocols. Patients undergone RBS during 2016-2020 will be considered a control group. The study will not involve any modification of the usual protocols. Statistical analyze: to make qualitative quantitative comparison regarding clinical and anthropometric factors between the two study groups (2021-22; 2016-20), the z-test for two proportions and t-test (two-tailed) will be used, respectively. The significance is fixed at 0.05 and all analyzes will be performed with the SPSS v.27 software. Expected results: enroll about 500 patients to obtain information on the safety of RBS and the current trends in Italy.

DETAILED DESCRIPTION:
Bariatric surgery is the most effective treatment for achieving significant long-term weight reduction and resolution of comorbidities, including diabetes mellitus, arterial hypertension, sleep apnea syndrome [1]. Revisional bariatric surgery (RBS) is an option for patients who have an inadequate response after bariatric surgery for weight loss and improvement/resolution of comorbidities, or significant weight regain after a satisfactory, initial response, even with comorbidities' relapse [2,3]. All bariatric procedures are subject to failure, in different proportions, based on the type and mechanism of action and the patient's compliance to follow-up. Recent studies suggest that revision rates for sleeve gastrectomy, which is the most performed bariatric surgery in the world since 2015 [4], can be as high as 10% when patients are followed for more than 3 years and as high as 22%. after 10 years [5].

Revisional bariatric surgery is a constantly growing set of procedures. The choice of the revision procedure must consider the indication, the primary technique, and the patient's characteristics [3,6-9]. There is a lack of high-quality studies and an almost total lack of randomized data [6] on various aspects of RBS. These factors make it difficult for individual surgeons treating these patients to know which RBS procedures to recommend to their patients, not least because there are no guidelines for choosing RBS [7].

As defined by the American Society for Metabolic and Bariatric Surgery (ASMBS) Revision Task Force, RBS includes conversion (procedures that change from one initial procedure to a different type), correction (procedures that address complications), and reversal (procedures that restore the original anatomy) [10].

RBS results in higher mortality and complication rates than primary procedures [5,6,11]. However, the literature reports an increasing trend in the percentage of "conversion" intent revision surgeries for IWL or WR based on self-referencing surgical center choices, in the absence of solid outcome data [3]. There is a lack of Italian data documenting the trend of RBS in the last 5 years (% of interventions for high-volume centers), the indications for "conversion", types of intervention and, above all, data on mortality and postoperative complications, essential for the informed consent offered to the patient candidate to RBS.

PRIMARY AIM: To analyze the trend, mortality, and complications at 30 days. SECONDARY AIMS: 30-day readmission rate, reoperations for any reason related to bariatric surgery.

Study's design: longitudinal, prospective, multicenter study. Time interval: 10 months (1 month of preparation and enrollment October 2021, 6 months of treatment November 2022 - April 2022, 1 month of follow-up May 2022, 4 months of data collection and analysis, manuscript preparation and publication May - July 2022).

Location: 11 high-volume bariatric centers of the Italian National Health Service (SSN), university hospitals, hospitals, accredited private centers.

METHODS: All bariatric revisional cases operated from 01.11.2021 - 31.04.2022 will be collected in a prospective, online database, within a dedicated website. Will be analyzed: indications; revision technique; mortality; intraoperative complications; perioperative complications; readmission to the hospital after discharge, for any reason.

All participating centers will follow the usual preoperative work-up protocol, surgical indication, informed consent, preparation for surgery and postoperative follow-up. No insurance is needed for this study, as it is an observation of routine clinical practice.

The patients operated on during the 2016-2020 period, in the same semester (November-April) will be considered as a comparative group (control group).

The prospective observational study will not involve any modification of the protocols in use in the individual centers.

Statistical analysis: categorical data will be described by absolute and relative frequency, continuous data by mean, standard deviation, and range. To make qualitative quantitative comparison regarding clinical and anthropometric factors between the two study groups (2021-22; 2016-20), the z-test for two proportions and t-test (two-tailed) will be used, respectively. The significance is fixed at 0.05 and all analyzes will be performed with the SPSS v.27 software. An online platform dedicated to the study for data entry will be used, as per the data collection form (CRF).

The study will be conducted in accordance with the principles of Good Clinical Practice, as well as with the study's protocol under registration within clinicaltrials.gov.

EXPECTED RESULTS: to enroll about 500 patients to obtain information on the safety of RBS and the current trend in Italy. DISCLOSURES: No funding is required or needed for this study. Researchers have nothing to reveal.

ELIGIBILITY:
Inclusion Criteria:

1. Previous bariatric surgery;
2. Age:> 18 <65 years;
3. Compensated comorbidities;
4. Official surgical informed consent with Covid-19 addendum in case the state of emergency continues.
5. Revisional bariatric procedures approved by: SICOB (Italian Society of Obesity Surgery), EAES (European Association for Endoscopic Surgery) and IFSO (International Federation for Obesity Surgery), including: Roux-en-Y gastric bypass, sleeve gastrectomy or repeated sleeve gastrectomy, biliopancreatic diversion, duodenal switch, duodenal-jejunal bypass, one-anastomosis gastric bypass, single anastomosis duodeno-ileal bypass (SAID), performed exclusively laparoscopically.

Routine performance expected during the clinical study, as inclusion criteria:

* obtaining the informed consent for participating in the clinical study;
* delivery of the privacy, information and data treatment forms;
* online data collection form's compilation (CRF);
* collection of specific Italian Society of Obesity Surgery (SICOB) informed consent for revisional bariatric surgery, COVID-19 regional questionnaire and SICOB's addendum for bariatric surgery during COVID-19 (attachment 6);
* emission of patients' letter of discharge, indicating the telephone interview after 7 and 15 days and the first outpatient check-up after 30 days;
* information letter for the general practitioner (see attachment 7);

Exclusion Criteria:

* no compliance to the inclusion criteria;
* other revisional bariatric procedures than ones approved;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group A: all consecutive patients undergoing RBS between November 2021 - April 2022 in all involved centers; Group B (control): all patients operated on for RBS during the 2016-2020 period, in the same semester (November - April) in all involved centers will be considered as a comparative group.
  All data will be collected anonymously, on a prospective, online database, with a dedicated website. Each centre will have its own slot for data submission like anthropometrics and date of primary BS, weight loss evolution, and reasons, date and anthropometrics for RBS, as well as 30-day postoperative evolution. The prospective observational study will not involve any major modification of the already established protocols, in use in each individual centers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | first 30 postoperative days
  Mortality after revisional bariatric surgery
Complications | first 30 postoperative days
  complications after revisional bariatric surgery

SECONDARY OUTCOMES:
Readmission | first 30 postoperative days
  readmission after revisional bariatric surgery
Reoperations | first 30 postoperative days
  reoperations for any reason related to revisional bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Silecchia, MD, PhD, Principal Investigator — Sapienza University of Rome, Italy
Locations (11):
- Italy (11):
  - UOC Chirurgia Generale, Ospedale Villa d'Agri, Potenza, Basilicate
  - University La Sapienza of Rome, Department of Medico-Surgical Sciences and Biotechnologies, Latina, LT
  - UOSD Week Surgery, Chirurgia Bariatrica, Azienda Ospedale-Università di Padova, Padua, Veneto
  - Policlinico San Marco, Istituti Ospedalieri Bergamaschi, GSD, Bergamo
  - UO Chirurgia Generale, Policlinico San Marco, Istituti Ospedalieri Bergamaschi, GSD, Bergamo
  - Unita di Chirurgia dell'Obesità e Metabolica, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Centre for the Study and Research of Treatment for Morbid Obesity, Department of Medical and Surgical Sciences, Alma Mater Studiorum University of Bologna,, Bologna
  - UOC di Chirurgia Generale e d'Urgenza, Presidio Ospedaliero ARNAS Garibaldi Nesima, Catania
  - UO di Chirurgia Bariatrica, Humanitas Research Hospital, Rozzano, Milan
  - UOC di Chirurgia Bariatrica e Metabolica, Azienda Ospedaliera Universitaria Pisana, Presidio Ospedaliero "Nuovo Santa Chiara", Pisa
  - UOC Chirurgia Bariatrica e Metabolica, Ospedale San Carlo di Nancy e Universita ''Tor Vergata" di Roma, Roma
  - Dipartimento di Scienze Chirurgiche, Azienda Ospedaliera Universitaria Città della Salute e della Scienza, Università di Torino, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stefanidis D, Malireddy K, Kuwada T, Phillips R, Zoog E, Gersin KS. Revisional bariatric surgery: perioperative morbidity is determined by type of procedure. Surg Endosc. 2013 Dec;27(12):4504-10. doi: 10.1007/s00464-013-3097-y. Epub 2013 Aug 14. PMID 23943144
- [Result] Mahawar KK, Himpens JM, Shikora SA, Ramos AC, Torres A, Somers S, Dillemans B, Angrisani L, Greve JWM, Chevallier JM, Chowbey P, De Luca M, Weiner R, Prager G, Vilallonga R, Adamo M, Sakran N, Kow L, Lakdawala M, Dargent J, Nimeri A, Small PK. The first consensus statement on revisional bariatric surgery using a modified Delphi approach. Surg Endosc. 2020 Apr;34(4):1648-1657. doi: 10.1007/s00464-019-06937-1. Epub 2019 Jun 19. PMID 31218425
- [Result] Angrisani L, Santonicola A, Iovino P, Vitiello A, Higa K, Himpens J, Buchwald H, Scopinaro N. IFSO Worldwide Survey 2016: Primary, Endoluminal, and Revisional Procedures. Obes Surg. 2018 Dec;28(12):3783-3794. doi: 10.1007/s11695-018-3450-2. PMID 30121858
- [Result] Guan B, Chong TH, Peng J, Chen Y, Wang C, Yang J. Mid-long-term Revisional Surgery After Sleeve Gastrectomy: a Systematic Review and Meta-analysis. Obes Surg. 2019 Jun;29(6):1965-1975. doi: 10.1007/s11695-019-03842-3. PMID 30903425
- [Result] Athanasiadis DI, Martin A, Kapsampelis P, Monfared S, Stefanidis D. Factors associated with weight regain post-bariatric surgery: a systematic review. Surg Endosc. 2021 Aug;35(8):4069-4084. doi: 10.1007/s00464-021-08329-w. Epub 2021 Mar 1. PMID 33650001
- [Result] Li S, Jiao S, Zhang S, Zhou J. Revisional Surgeries of Laparoscopic Sleeve Gastrectomy. Diabetes Metab Syndr Obes. 2021 Feb 10;14:575-588. doi: 10.2147/DMSO.S295162. eCollection 2021. PMID 33603423
- [Result] Di Lorenzo N, Antoniou SA, Batterham RL, Busetto L, Godoroja D, Iossa A, Carrano FM, Agresta F, Alarcon I, Azran C, Bouvy N, Balague Ponz C, Buza M, Copaescu C, De Luca M, Dicker D, Di Vincenzo A, Felsenreich DM, Francis NK, Fried M, Gonzalo Prats B, Goitein D, Halford JCG, Herlesova J, Kalogridaki M, Ket H, Morales-Conde S, Piatto G, Prager G, Pruijssers S, Pucci A, Rayman S, Romano E, Sanchez-Cordero S, Vilallonga R, Silecchia G. Clinical practice guidelines of the European Association for Endoscopic Surgery (EAES) on bariatric surgery: update 2020 endorsed by IFSO-EC, EASO and ESPCOP. Surg Endosc. 2020 Jun;34(6):2332-2358. doi: 10.1007/s00464-020-07555-y. Epub 2020 Apr 23. PMID 32328827
- [Result] Radtka JF 3rd, Puleo FJ, Wang L, Cooney RN. Revisional bariatric surgery: who, what, where, and when? Surg Obes Relat Dis. 2010 Nov-Dec;6(6):635-42. doi: 10.1016/j.soard.2010.04.005. Epub 2010 May 4. PMID 20702147
- [Result] Kellogg TA. Revisional bariatric surgery. Surg Clin North Am. 2011 Dec;91(6):1353-71, x. doi: 10.1016/j.suc.2011.08.004. PMID 22054158
- [Result] Brolin RE, Cody RP. Weight loss outcome of revisional bariatric operations varies according to the primary procedure. Ann Surg. 2008 Aug;248(2):227-32. doi: 10.1097/SLA.0b013e3181820cdf. PMID 18650632
- [Result] Brethauer SA, Kothari S, Sudan R, Williams B, English WJ, Brengman M, Kurian M, Hutter M, Stegemann L, Kallies K, Nguyen NT, Ponce J, Morton JM. Systematic review on reoperative bariatric surgery: American Society for Metabolic and Bariatric Surgery Revision Task Force. Surg Obes Relat Dis. 2014 Sep-Oct;10(5):952-72. doi: 10.1016/j.soard.2014.02.014. Epub 2014 Feb 22. PMID 24776071
- [Result] Abdelgawad M, De Angelis F, Iossa A, Rizzello M, Cavallaro G, Silecchia G. Management of Complications and Outcomes After Revisional Bariatric Surgery: 3-Year Experience at a Bariatric Center of Excellence. Obes Surg. 2016 Sep;26(9):2144-2149. doi: 10.1007/s11695-016-2071-x. PMID 26809671
- [Result] Koh ZJ, Chew CAZ, Zhang JJY, Syn N, Kim G, Yan So JB, Shabbir A. Metabolic outcomes after revisional bariatric surgery: a systematic review and meta-analysis. Surg Obes Relat Dis. 2020 Oct;16(10):1442-1454. doi: 10.1016/j.soard.2020.05.029. Epub 2020 Jun 6. PMID 32711955
- [Result] Boru CE, Greco F, Giustacchini P, Raffaelli M, Silecchia G. Short-term outcomes of sleeve gastrectomy conversion to R-Y gastric bypass: multi-center retrospective study. Langenbecks Arch Surg. 2018 Jun;403(4):473-479. doi: 10.1007/s00423-018-1675-0. Epub 2018 Apr 20. PMID 29675614
- [Result] Vilallonga R, Fort JM, Rodriguez Luna MR, Garcia Ruiz de Gordejuela A, Gonzalez O, Caubet E, Cirera de Tudela A, Palermo M, Ciudin A, Armengol M. The Panoramic View of Revisional Bariatric Surgery. J Laparoendosc Adv Surg Tech A. 2021 Sep 6. doi: 10.1089/lap.2021.0506. Online ahead of print. PMID 34492201
- [Result] Palermo M, Khwaja H. Overview of Revisional Bariatric Surgery. J Laparoendosc Adv Surg Tech A. 2021 Sep 6. doi: 10.1089/lap.2021.0554. Online ahead of print. No abstract available. PMID 34491846
- [Result] Akpinar EO, Marang-van de Mheen PJ, Nienhuijs SW, Greve JWM, Liem RSL. National Bariatric Surgery Registries: an International Comparison. Obes Surg. 2021 Jul;31(7):3031-3039. doi: 10.1007/s11695-021-05359-0. Epub 2021 Mar 30. PMID 33786743